CLINICAL TRIAL: NCT02594644
Title: The Use of Microneedles to Expedite Treatment Time in Photodynamic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 553703
Record Dates: First submitted 2015-10-31; First posted 2015-11-03 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-10

CONDITIONS: Keratosis, Actinic
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Blue Light

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10-minute Incubation with Microneedle Roller & Sham (Experimental): 10-minute topical aminolevulinic acid incubation group. Subjects randomized by binary randomization into each treatment group and undergo secondary binary randomization for microneedle roller treatment (vs. sham microneedle) to the right or left side of the face. Blue light therapy follows.
  Interventions: Device: Microneedle Roller; Drug: Aminolevulinic Acid; Radiation: Blue Light
- 20-minute Incubation with Microneedle Roller & Sham (Experimental): 20-minute topical aminolevulinic acid incubation group. Subjects randomized by binary randomization into each treatment group and undergo secondary binary randomization for microneedle roller treatment (vs. sham microneedle) to the right or left side of the face. Blue light therapy follows.
  Interventions: Device: Microneedle Roller; Drug: Aminolevulinic Acid; Radiation: Blue Light

INTERVENTIONS:
Device: Microneedle Roller — The study device (MR200, Clinical Resolutions Laboratory, Inc.) is a disposable roller equipped with stainless steel needles that are 650 micrometers in length.
Drug: Aminolevulinic Acid — Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
Radiation: Blue Light — Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA

SUMMARY:
The aim of this study is to investigate how varying incubation periods of topical aminolevulinic acid after pretreatment with microneedle application can facilitate the penetration and efficacy of photodynamic therapy.

DETAILED DESCRIPTION:
The current standard of care of photodynamic therapy to treat actinic keratoses includes pre-treatment of the area with topical aminolevulinic acid for 1 hour, followed by treatment with blue light. In a previous study, the investigators showed pretreatment of microneedles enhance penetration of topical aminolevulinic acid as compared to the control group.

The aim of this study is to investigate how varying incubation periods of topical aminolevulinic acid after pretreatment with microneedle application can facilitate the penetration and efficacy of photodynamic therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Subjects has actinic keratoses and qualifies for photodynamic therapy
* Do not meet any of the exclusion criteria

Exclusion Criteria:

* Subjects who smoke
* Subjects who have a photosensitizing condition such as lupus, porphyria, or similar condition
* Subjects who have established allergy to topical ALA
* Subjects who have had a documented nonmelanoma skin cancer on the face over the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2016-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California-Davis, Department of Dermatology, Sacramento, California, United States

REFERENCES:
- [Derived] Petukhova TA, Hassoun LA, Foolad N, Barath M, Sivamani RK. Effect of Expedited Microneedle-Assisted Photodynamic Therapy for Field Treatment of Actinic Keratoses: A Randomized Clinical Trial. JAMA Dermatol. 2017 Jul 1;153(7):637-643. doi: 10.1001/jamadermatol.2017.0849. PMID 28514458

RESULTS

PARTICIPANT FLOW:
Groups:
- 10-minute Incubation With Microneedle Roller & Sham: 10-minute topical aminolevulinic acid incubation group. Subjects randomized by binary randomization into each treatment group and undergo secondary binary randomization for microneedle roller treatment (vs. sham microneedle) to the right or left side of the face. Blue light therapy follows.
  Microneedle Roller: The study device (MR200, Clinical Resolutions Laboratory, Inc.) is a disposable roller equipped with stainless steel needles that are 200 micrometers in length.
  Aminolevulinic Acid: Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
  Blue Light: Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA
- 20-minute Incubation With Microneedle Roller: 20-minute topical aminolevulinic acid incubation group. Subjects randomized by binary randomization into each treatment group and undergo secondary binary randomization for microneedle roller treatment (vs. sham microneedle) to the right or left side of the face. Blue light therapy follows.
  Microneedle Roller: The study device (MR200, Clinical Resolutions Laboratory, Inc.) is a disposable roller equipped with stainless steel needles that are 200 micrometers in length.
  Aminolevulinic Acid: Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
  Blue Light: Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA
Period: Overall Study
Arm/Group | 10-minute Incubation With Microneedle Roller & Sham | 20-minute Incubation With Microneedle Roller
Started | 16 | 16
Completed | 16 | 15
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: In each group we initially enrolled 16 participants. In the 20 minute incubation group, we had 1 dropout which left us with 15 participants that finished.
Groups:
- 20-minute Incubation With Microneedle Roller & Sham: 20-minute topical aminolevulinic acid incubation group. Subjects randomized by binary randomization into each treatment group and undergo secondary binary randomization for microneedle roller treatment (vs. sham microneedle) to the right or left side of the face. Blue light therapy follows.
  Microneedle Roller: The study device (MR200, Clinical Resolutions Laboratory, Inc.) is a disposable roller equipped with stainless steel needles that are 200 micrometers in length.
  Aminolevulinic Acid: Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
  Blue Light: Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA
- Total: Total of all reporting groups
Arm/Group | 10-minute Incubation With Microneedle Roller & Sham | 20-minute Incubation With Microneedle Roller & Sham | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 15
  >=65 years | 11 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4375 (9.858795) | 62.75 (8.575158) | 64.09 (9.19101)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 11 | 11 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Percentage of Complete Clearance of the Actinic Keratoses
Description: The primary endpoint will be the difference in the percentage of complete clearance of the actinic keratoses as an intraindividual comparison between the treatment groups.
Time Frame: Baseline, 2 Months
Measure: Mean (Standard Error); unit: Percentage of AK Clearance
Groups:
- 10-minute Incubation With Microneedle Roller: 10-minute topical aminolevulinic acid incubation group. Subjects randomized by binary randomization into each treatment group and undergo secondary binary randomization for microneedle roller treatment (vs. sham microneedle) to the right or left side of the face. Blue light therapy follows.
  Microneedle Roller: The study device (MR200, Clinical Resolutions Laboratory, Inc.) is a disposable roller equipped with stainless steel needles that are 200 micrometers in length.
  Aminolevulinic Acid: Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
  Blue Light: Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA
- 10-minute Incubation With Sham Microneedles: 10-minute topical aminolevulinic acid incubation group. Binary randomization of subjects into treatment groups and secondary binary randomization for application of the microneedle roller treatment (vs. sham microneedle) to the right or left side of the face. Blue light therapy follows.
  Aminolevulinic Acid: Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
  Blue Light: Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA
- 20-minute Incubation With Sham Microneedles: 20-minute topical aminolevulinic acid incubation group. Binary randomization of subjects into treatment groups and secondary binary randomization for application of the microneedle roller treatment (vs. sham microneedle) to the right or left side of the face. Blue light therapy follows.
  Aminolevulinic Acid: Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
  Blue Light: Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA
Arm/Group | 10-minute Incubation With Microneedle Roller | 20-minute Incubation With Microneedle Roller | 10-minute Incubation With Sham Microneedles | 20-minute Incubation With Sham Microneedles
Number analyzed (Participants) | 16 | 16 | 16 | 16
Percentage of AK Clearance | 43 (13) | 76 (3.9) | 38 (8.1) | 58 (5.7)

2. Secondary Outcome: Visual Analog Pain Scale
Description: The secondary will be any pain associated with the microneedle pretreatment and with the application of the PDT using the 100 mm Visual Analog Scale pain grading. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Time Frame: Immediately Post-Treatment
Measure: Mean (Standard Error); unit: Millimeters
Groups:
- Pain_microneedle: 10-minute Incubation With Microneedle Roller; Pain_microneedle: 10-minute Incubation With Microneedle Sham; Pain_PDT: 10-minute Incubation With Microneedle Sham; Pain_PDT: 10-minute Incubation With Microneedle Roller: 10-minute topical aminolevulinic acid incubation group. Subjects randomized by binary randomization into each treatment group and undergo secondary binary randomization for microneedle roller treatment (vs. sham microneedle) to the right or left side of the face. Blue light therapy follows.
  Microneedle Roller: The study device (MR200, Clinical Resolutions Laboratory, Inc.) is a disposable roller equipped with stainless steel needles that are 200 micrometers in length.
  Aminolevulinic Acid: Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
  Blue Light: Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA
- Pain_microneedle: 20-minute Incubation With Microneedle Roller; Pain_microneedle: 20-minute Incubation With Microneedle Sham; Pain_PDT: 20-minute Incubation With Microneedle Sham; Pain_PDT: 20-minute Incubation With Microneedle Roller: 20-minute topical aminolevulinic acid incubation group. Subjects randomized by binary randomization into each treatment group and undergo secondary binary randomization for microneedle roller treatment (vs. sham microneedle) to the right or left side of the face. Blue light therapy follows.
  Microneedle Roller: The study device (MR200, Clinical Resolutions Laboratory, Inc.) is a disposable roller equipped with stainless steel needles that are 200 micrometers in length.
  Aminolevulinic Acid: Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
  Blue Light: Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA
Arm/Group | Pain_microneedle: 10-minute Incubation With Microneedle Roller | Pain_microneedle: 20-minute Incubation With Microneedle Roller | Pain_microneedle: 10-minute Incubation With Microneedle Sham | Pain_microneedle: 20-minute Incubation With Microneedle Sham | Pain_PDT: 10-minute Incubation With Microneedle Sham | Pain_PDT: 10-minute Incubation With Microneedle Roller | Pain_PDT: 20-minute Incubation With Microneedle Sham | Pain_PDT: 20-minute Incubation With Microneedle Roller
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16
Millimeters | 1.4 (.5) | 1.3 (.4) | .3 (.2) | .3 (.2) | 0.3 (0.2) | .5 (.2) | 0.4 (0.1) | .7 (.2)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | 10-minute Incubation With Microneedle Roller & Sham | 20-minute Incubation With Microneedle Roller & Sham
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No